CLINICAL TRIAL: NCT07193797
Title: Clinical Phenotypes of ICU Delirium and Subsequent Impairment of Physical, Cognitive and Mental Health During Transition From ICU to Hospital Wards
Brief Title: Delirium Phenotypes and Subsequent Impairment During Transition From ICU to Hospital Wards
Status: Recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Sponsor
Other Study IDs: NSFC-7220040527
Record Dates: First submitted 2025-01-12; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-01

CONDITIONS: Delirium; Post ICU Syndrome
Keywords: ICU delirium; Phenotypes; Physical impairment; Cognitive impairment; Mental health impairment; ICU transition
MeSH Terms: conditions — Delirium; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICU delirium cohort
  Interventions: Other: Phenotypes of ICU delirium

INTERVENTIONS:
Other: Phenotypes of ICU delirium — The included delirium patients will be divided into different phenotypes, according to delirium risk factors such as age, history of cerebrovascular accident, blood transfusion, surgery duration etc.

SUMMARY:
The goal of this observational study is to learn about the disability profile during transition from ICU to hospital wards of delirium patients, including cognitive impairment, physical dysfunction and psychological disorders. The main question it aims to answer is:

* What is the main rehabilitation problem during transition from ICU to hospital wards for patients who experienced ICU delirium?
* Dose different phenotypes of ICU delirium shows different rehabilitation problem during ICU transition? Participants will be followed up and assessed by questionnaires after discharge from ICU to hospital wards until hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* patients aged above 18-year-old
* at least one positive screening of CAM-ICU (Confusion Assessment Method for ICU) assessment during ICU stay
* patients are transferred to hospital ward after ICU discharge

Exclusion Criteria:

* patients are with severe dementia
* blindness, deafness or inability to understand mandarin
* life expectancy of less than 24h
* stayed in ICU more than one-month after the first CAM-ICU positive screening

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to ICU and developed delirium will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 189 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Physical impairment | At first, third day and fifth day after ICU discharge, at the 1 day of hospital discharge, one-month after hospital discharge
  The Modified Barthel Index is a widely used scale for assessing a patient's level of independence in activities of daily living (ADLs). Each activity is scored based on the degree of assistance required, with total scores typically ranging from 0 (complete dependence) to 100 (complete independence).
Cognitive impairment | At first, third day and fifth day after ICU discharge, at the 1 day of hospital discharge, one-month after hospital discharge
  The Mini-MoCA (Mini Montreal Cognitive Assessment) is a brief cognitive screening tool derived from the full MoCA, designed to rapidly assess cognitive function in clinical and hospital settings. It evaluates key domains such as orientation, attention, memory, language, and visuospatial skills, using a condensed format suitable for bedside.
Mental health | At first, third day and fifth day after ICU discharge, at the 1 day of hospital discharge, one-month after hospital discharge
  Hospital Anxiety and Depression Scale(HADS) is a 14-item tool used to screen for anxiety and depression in hospitalised patients. It includes two 7-item subscales, each scored 0-21, with higher scores indicate more severe psychological distress.

SECONDARY OUTCOMES:
Hospital stay | up to 30 days
  Duration of hospital stay
In-hospital Mortality | up to 30 days
  Mortality during hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No